CLINICAL TRIAL: NCT07278726
Title: Upfront Targeted Axillary Dissection for Luminal Breast Cancer With Limited Axillary Involvement: the UTAD Study of the Italian National Association of Breast Surgeons (ANISC)
Brief Title: Upfront Targeted Axillary Dissection for Luminal Breast Cancer With Limited Axillary Involvement
Acronym: UTAD
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 5132; L2-439 (Other: Comitato Etico Territoriale Lombardia 2)
Record Dates: First submitted 2025-11-17; First posted 2025-12-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: ALND; Sentinel Lymph Node Biopsy (SLNB); Targeted Axillary Dissection (TAD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Upfront Targeted Axillary Dissection (UTAD) — During the surgical intervention lymphnodes excised both with reflector localization and Gamma probe will be sent for pathological examination and only in case of more than 2 metastatic lymph nodes (and at least one of them with macrometastasis) axillary dissection will be performed.

SUMMARY:
The present study aims to avoid axillary lymph node dissection (ALND) in patients with an Ultrasound (US) detected positive preoperative lymph node involvement (1 or 2 suspicious lymph-nodes) and a needle histology/cytology placing a marker in the most suspicious node undergoing upfront surgery if neoadjuvant treatment is not indicated. The marked lymph node will be retrieved along with sentinel lymphnode(SLN)(s) to minimize the false-negative rate and only in case of ≥3 positive SLNs ALND will be performed, in order to minimize surgical overtreatment among women with preoperatively confirmed axillary nodal metastasis.

DETAILED DESCRIPTION:
The patients that will avoid axillary lymph node dissection (ALND) meet all the criteria listed in the latest NCCN guidelines version.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T0-T1-T2 ER+/PR+ HER2- breast cancer with limited nodal involvement (1 or 2 suspicious lymph node on US, with at least 1 nodal positive cytology/histology)
* M0
* Conservative surgery or mastectomy
* Neoadjuvant treatment not recommended after a multidisciplinary discussion
* Patients between 18 and 90 years old
* Patients willing and able to follow the study procedures and available for follow-up over the entire duration of the study

Exclusion Criteria:

* Psychiatric, addictive or any disorder, which compromises ability to give informed consent for participation in the study
* Personal history of invasive breast cancer
* Other invasive malignancies diagnosed in the last five years
* Any condition that may expose the individual to a higher risk or preclude the study from achieving full compliance or completion
* Contraindications to radiation therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with T0-T1-T2 ER+ HER2- breast cancer with limited nodal involvement (1 or 2 suspicious lymph node on US, with at least 1 positive nodal citology/histology) M0 for whom neoadjuvant treatment is not recommended after a multidisciplinary discussion, between 18 and 90 years old willing and able to follow the study procedures and available for follow-up over the entire duration of the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2033-11 (Estimated)

PRIMARY OUTCOMES:
Successful rate of the retrieval of the deflector. | Perioperative/Periprocedural
  Number of successful retrieval of the deflector on the total number of surgeries.
Prevention of Axillary Lymph Node Dissection | Perioperative/Periprocedural
  Total number of patient that did not received but were elegible for Axillary Lymph Node Dissection by the current guidelines on the total number of surgeries.

SECONDARY OUTCOMES:
Axillary recurrence rate | 5 years from surgery.
  The secondary endpoint is the rate of axillary recurrence in patients undergoing UTAD and who avoid AD. Cumulative incidence of axillary recurrence as first event will be calculated, considering the following events as competing: distant metastases, death, second primary malignancies, invasive ipsilateral tumor recurrences in the breast or chest wall, supraclavicular or internal mammary recurrences, and contralateral invasive cancers.

CONTACTS AND LOCATIONS:
Locations (14):
- Italy (13):
  - IRCCS AOU di Bologna - Policlinico di Sant'Orsola, Bologna, Italy
  - AUSL Romagna - Presidio Ospedaliero Morgagni-Pierantoni, Forlì, Italy
  - European Institute of Oncology, Milan, Italy
  - Fondazione IRCCS Istituto Nazionale Tumori di Milano, Milan, Italy
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Italy
  - Presidio Ospedaliero "G. Bernabeo", Ortona, Italy
  - Policlinico San Matteo, Pavia, Italy
  - Azienda Ospedaliera Universitaria Pisana, Pisa, Italy
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy
  - AO San Giovanni Addolorata, Roma, Italy
  - IRCCS Humanitas Research Hospital, Rozzano, Italy
  - Azienda sanitaria universitaria Giuliano Isontina, Trieste, Italy
  - ASST Sette Laghi - Ospedale di Circolo e Fondazione Macchi, Varese, Italy
- Ente Ospedaliero Cantonale, Lugano, Switzerland, Switzerland

IPD SHARING:
Plan to Share IPD: No